CLINICAL TRIAL: NCT06335849
Title: A Phase I, Randomized, Observer-blinded, Positive-Controlled, Dose Escalation Clinical Trial to Assess the Safety and Immunogenicity of the Recombinant Zoster Vaccine （CHO Cell）, LYB004 in Adults Aged 50 to 70 Years
Brief Title: A Safety and Immunogenicity Trial of the Recombinant Zoster Vaccine （CHO Cell）, LYB004 in Adults Aged 50 to 70 Years
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Guangzhou Patronus Biotech Co., Ltd. (Industry)
Collaborators: Yantai Patronus Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LYB004-CT-AUS-101
Record Dates: First submitted 2024-03-13; First posted 2024-03-28 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Herpes Zoster
Keywords: Recombinant Zoster Vaccine; Glycoprotein E; Varicella-Zoster Virus; Herpes zoster; Shingles
MeSH Terms: conditions — Herpes Zoster; Chickenpox

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Treatment 1 (LYB004 25µg) (Experimental): Subjects will be enrolled and stratified by age (50-59 years and 60-70 years in a 1:1 ratio) and randomized (2:2:1) to receive 25 μg LYB004, 50 μg LYB004 or SHINGRIX. The two-dose immunization schedule will be adopted, that is, LYB004 or SHINGRIX will be intramuscularly injected on Day 0 and Day 60.
  Interventions: Biological: LYB004 25µg
- Treatment 2 (LYB004 50µg) (Experimental): Subjects will be enrolled and stratified by age (50-59 years and 60-70 years in a 1:1 ratio) and randomized (2:2:1) to receive 25 μg LYB004, 50 μg LYB004 or SHINGRIX. The two-dose immunization schedule will be adopted, that is, LYB004 or SHINGRIX will be intramuscularly injected on Day 0 and Day 60.
  Interventions: Biological: LYB004 50µg
- Treatment 3 (SHINGRIX) (Active Comparator): Subjects will be enrolled and stratified by age (50-59 years and 60-70 years in a 1:1 ratio) and randomized (2:2:1) to receive 25 μg LYB004, 50 μg LYB004 or SHINGRIX. The two-dose immunization schedule will be adopted, that is, LYB004 or SHINGRIX will be intramuscularly injected on Day 0 and Day 60.
  Interventions: Biological: SHINGRIX

INTERVENTIONS:
Biological: LYB004 25µg — Subjects will be enrolled and stratified by age (50-59 years and 60-70 years in a 1:1 ratio) and randomized (2:2:1) to receive 25 μg LYB004, 50 μg LYB004 or SHINGRIX. The two-dose immunization schedule will be adopted, that is, LYB004 or SHINGRIX will be intramuscularly injected on Day 0 and Day 60.
  Arms: Treatment 1 (LYB004 25µg)
Biological: LYB004 50µg — Subjects will be enrolled and stratified by age (50-59 years and 60-70 years in a 1:1 ratio) and randomized (2:2:1) to receive 25 μg LYB004, 50 μg LYB004 or SHINGRIX. The two-dose immunization schedule will be adopted, that is, LYB004 or SHINGRIX will be intramuscularly injected on Day 0 and Day 60.
  Arms: Treatment 2 (LYB004 50µg)
Biological: SHINGRIX — Subjects will be enrolled and stratified by age (50-59 years and 60-70 years in a 1:1 ratio) and randomized (2:2:1) to receive 25 μg LYB004, 50 μg LYB004 or SHINGRIX. The two-dose immunization schedule will be adopted, that is, LYB004 or SHINGRIX will be intramuscularly injected on Day 0 and Day 60.
  Arms: Treatment 3 (SHINGRIX)

SUMMARY:
This phase 1 study in Australia will evaluate the safety and immunogenicity of the Recombinant Zoster Vaccine (CHO Cell), LYB004 in Adults Aged 50 to 70 Years.

DETAILED DESCRIPTION:
A randomized, observer-blinded, positive-controlled, dose escalation trial will be conducted to observe the safety and immunogenicity of LYB004 in adults 50 to 70 years of age. A total of 48 healthy subjects will be enrolled and stratified by age (50-59 years and 60-70 years in a 1:1 ratio) and randomized (2:1) to receive LYB004 or SHINGRIX. Two dose levels of LYB004 will be provided, low dose 25 μg and high dose 50 μg. The two-dose immunization schedule will be adopted, that is, LYB004 or SHINGRIX will be intramuscularly injected on Day 0 and Day 60, respectively.

ELIGIBILITY:
Inclusion Criteria:

1. A male or female aged 50 to 70 years inclusive at screening.
2. Written informed consent obtained from the subject before any assessment is performed.
3. Subjects who the investigator believes that they can and will comply with the requirements of the protocol. (e.g., complete the diary cards, and complete follow-up visits).
4. Subjects must have a Body Mass Index (BMI) between ≥18.0 and ≤35.0 kg/m^2 at screening.
5. Female subjects who are not pregnant or lactating. Female subjects with childbearing potential and their partners should use highly effective, medically accepted double-barrier contraception and will not have pregnancy and fertility plan until study completion.

   * Female subjects of childbearing potential are defined as sexually mature women: 1) have not undergone hysterectomy, bilateral salpingectomy, and bilateral oophorectomy; 2) have had natural menses at any time in the preceding 12 consecutive months (without an alternative medical cause).
   * Highly effective double-barrier contraception is defined as use of a condom AND one of the following: Birth control pills (The Pill), Depot or injectable birth control, Intrauterine device (IUD), Birth Control Patch (e.g., Ortho Evra), NuvaRing®, Implantable contraception (e.g., Implanon).
6. Males participating in this study must agree to use highly effective, medically accepted double-barrier contraception (as described above) and refrain from donating sperm until study completion.

Exclusion Criteria:

1. Tympanic temperature > 37.5°C at screening.
2. History of HZ.
3. Previous vaccination against HZ or varicella. Planned administration of VZV or HZ vaccination during the study (including an investigational or non-registered vaccine), except for the investigational vaccine.
4. Received a live attenuated vaccine within 28 days before vaccination or received other vaccines within 14 days before vaccination.
5. Received any immunoglobulins or blood/plasma products within 3 months prior to vaccination.
6. Individuals with the following diseases: 1）Any acute disease or acute attack of chronic diseases or using antipyretic, analgesic or anti-allergic drugs (e.g., acetaminophen, ibuprofen, aspirin, loratadine, cetirizine, etc.) within 3 days prior to enrolment; 2）Allergies to any component of the investigational vaccine; 3）Subject has any clinically significant history of allergic conditions to other vaccines. 4）History of neurological disorders (convulsions, epilepsy, encephalopathy, etc.) or psychiatric disorders (bipolar disorder, schizophrenia, etc.) that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the participant inappropriate for entry into this study; 5）Asplenia, or functional asplenia; 6）Congenital or acquired immunodeficiency or autoimmune disease; 7）Chronic administration (≥14 consecutive days) of glucocorticoid (reference value for dose: ≥20 mg/day prednisone or equivalent) or other immunosuppressive agents within the past 3 months, with the exception of inhaled or topical steroids, or short-term use (<14 consecutive days) of oral corticosteroids; 8）Has severe cardiovascular diseases (cardiopulmonary disease, pulmonary edema), severe hepatic or renal diseases, and diabetes complications that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the participant inappropriate for entry into this study; 9）History of thrombocytopenia or other coagulation disorders which may be contraindications for an IM; 10）Severe hypertension uncontrolled by medication with systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥100 mmHg; 11）Positive test for Hepatitis C virus (HCV), Hepatitis B surface antigen (HbsAg), Human immunodeficiency virus (HIV) at screening; 12）Any skin condition and/or tattoo that may interfere with the evaluation of safety at the injection site.
7. Clinically significant laboratory abnormalities determined by the investigator prior to vaccination.
8. A positive urine drug test or alcohol breath test or a history of drug or alcohol abuse in the past 1 years.
9. Recent participation in another clinical trial, with receipt of the investigational drug/vaccine within 30 days prior to screening. Current participation or those planning to participate in another clinical trial during the study.
10. Other conditions that may impact the subject's safety or influence the assessment of vaccine response, as determined by the investigator.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-03-27 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate the reactogenicity of LYB004 vaccine | Within 30 minutes after each vaccination
  The incidence and severity of any adverse events (AEs) within 30 minutes after each vaccination
Evaluate the safety and reactogenicity of LYB004 vaccine | Within 0-7 days after each vaccination
  The incidence and severity of any solicited local and systemic AEs and unsolicited AEs within 0-7 days after each vaccination
Evaluate the safety of LYB004 vaccine | Within 30 days after each vaccination
  The incidence and severity of any AEs within 30 days after each vaccination
Evaluate the safety and tolerability in laboratory tests of LYB004 vaccine | 3 days, 14 days after each vaccination and 90 days after the first vaccination
  The occurrence of clinically significant laboratory abnormalities 3 days, 14 days after each vaccination and 90 days after the first vaccination
Evaluate the SAEs and AESIs of LYB004 vaccine | From the first vaccination up to 6 months after the second vaccination
  The incidence of any serious adverse events (SAEs) and adverse events of special interest (AESIs) from the first vaccination up to 6 months after the second vaccination

SECONDARY OUTCOMES:
Observe the humoral immunity of LYB004 vaccine | At 14 and 30 days after each vaccination
  The geometric mean concentration (GMC in mIU/ml), geometric mean fold rise (GMFR), and serum seroconversion rate (%) of gE antibodies at 14 and 30 days after each vaccination; the geometric mean titer (GMT in 1:X), GMFR, and serum seroconversion rate (%) of VZV antibodies at 14 and 30 days after each vaccination
Observe the cellular immunity of LYB004 vaccine | At 30 days after the second vaccination
  The frequency and the cell mediated immunity (CMI) response rate (%) of gE-specific CD4^2+ and CD8^2+ T cells (expressing at least 2 different activation markers: IFN-γ, IL-2, TNF-α, and CD40L) per 10^6 CD4 and CD8 T cells at 30 days after the second vaccination
Observe the persistence of humoral immunity of LYB004 vaccine | At 6 months after full vaccination
  The GMC in mIU/ml, GMFR, and serum seroconversion rate (%) of gE antibodies at 6 months after the second vaccination; the GMT in 1:X, GMFR, and serum seroconversion rate (%) of VZV antibodies at 6 months after the second vaccination
Observe the persistence of cellular immunity of LYB004 vaccine | At 6 months after full vaccination
  The frequency and the CMI response rate (%) of gE-specific CD4^2+ and CD8^2+T cells per 10^6 CD4 and CD8 T cells at 6 months after the second vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Christina Chang, M.D, Principal Investigator — Nucleus Network Pty Ltd.
Locations (1):
- Nucleus Network Pty Ltd, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No